CLINICAL TRIAL: NCT05995990
Title: Raman Spectral Imaging for Liver Tumours Following Liver Surgery
Brief Title: Raman Spectroscopy for Liver Tumours Following Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20ON038
Record Dates: First submitted 2021-07-23; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal liver metatases (Experimental): Liver tissue containing colorectal liver metastases
  Interventions: Device: Raman Spectrometry

INTERVENTIONS:
Device: Raman Spectrometry — Laboratory technique of Raman Spectrometry

SUMMARY:
The aim of the proposed research is to develop a quick and reliable method for automated evaluation of tissue sections for residual tumour in histology specimens following liver surgery. This advanced technology will enable assessment of liver tumours and resection margins following liver surgery. The technology is based on Raman spectroscopy (RS) and multivariate spectral analysis to produce 2-dimensional biochemical images that can reliably separate the spectral signal of liver tumours from surrounding normal tissue.

DETAILED DESCRIPTION:
In this proposal, investigators will investigate the ability of RS to distinguish between normal versus cancer in tissue blocks following liver surgery. If successful, this technique can then be investigated for intra-operative assessment efficacy to ensure that the resection margin of the tumour is clear (free of tumour cells), enabling this powerful procedure to be applied to all patients undergoing liver surgery for highest standard of care. This device is an early concept development of an In-Vitro Diagnostic Medical Device.

In this project investigators will answer the following two questions:

* Can Raman spectroscopy discriminate between healthy tissue and colorectal liver metastases? If yes, with what accuracy?
* How fast can a Raman spectroscopy image of a tissue section be built? The success of this research will lead to a significant improvement in the quality and efficiency of liver surgery for colorectal liver metastases as it will allow all patients undergoing surgery to benefit from the best treatment available to ensure resection margins are clear. Making the best techniques more widely available to all patients who need them reduces inequality in healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for liver tumours (colorectal liver metastases).
* Able to give informed consent.

Exclusion Criteria:

• Patients where there is any doubt regarding the diagnosis from pathologist as ascertained by previous diagnostic biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Raman spectroscopy is able to discriminate between healthy liver tissue and colorectal liver metastases. | 3 years
  To determine whether Raman spectroscopy can discriminate between healthy liver tissue and liver tumours.

SECONDARY OUTCOMES:
Tissue sections can be analysed by Raman spectroscopy more time effectively than normal clinical practice. | 3 years
  To determine how fast a Raman spectroscopy image of a tissue section can be built.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanwant Gomez, FRCS, Principal Investigator — Nottingham University Hospitals NHS Trust; Ioan Notingher, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Queens Medical Centre Campus, Nottingham, Nottinghamshire, United Kingdom